CLINICAL TRIAL: NCT00010959
Title: A Phase I Single-Dose Pharmacokinetic Study of Black Cohosh and Red Clover in Healthy Menopausal Women 45-59 Years of Age
Brief Title: Single-Dose Study of Black Cohosh and Red Clover
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); Office of Dietary Supplements (ODS) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P50AT000155-01P4 (NIH); P50AT000155-01 (NIH); NCT00008970 (obsolete NCT alias)
Record Dates: First submitted 2001-02-02; First posted 2001-02-05 (Estimated); Last update posted 2007-03-02 (Estimated); Status verified 2007-03

CONDITIONS: Menopause
Keywords: menopause; hot flashes; botanicals
MeSH Terms: conditions — Hot Flashes | interventions — black cohosh root extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cimicifuga racemosa
Drug: Trifolium pratense

SUMMARY:
This Phase I study will assess the pharmacokinetics of two botanicals, Trifolium pratense (red clover) and Cimicifuga racemosa (black cohosh). Participants will receive a single dose of one botanical preparation. The observation period will be one week. Drug toxicity, absorption, distribution, metabolism and elimination data will be collected, and dosages to be utilized in a Phase II clinical trial will be determined.

DETAILED DESCRIPTION:
This Phase I study will assess the pharmacokinetics of two botanicals, Trifolium pratense (red clover) and Cimicifuga racemosa (black cohosh). Participants will receive a single dose of one botanical preparation. The observation period will be one week. Drug toxicity, absorption, distribution, metabolism and elimination data will be collected, and dosages to be utilized in a Phase II clinical trial will be determined. The Phase II trial will examine the efficacies of red clover and black cohosh for the reduction of menopausal symptoms in healthy menopausal women. The study will be randomized, double-blinded, and placebo-controlled. Study duration will be one year.

ELIGIBILITY:
Inclusion Criteria:

* Healthy menopausal women
* Average body weight
* Able to give informed consent

Exclusion Criteria:

* Smoker
* Use of any prescription medicine within the last 2 months
* Obesity > 30% above ideal body weight
* Previous history of breast or reproductive cancer
* Alcohol abuse or consumption above 5 glasses of wine per week or equivalent
* Chronic disease such as diabetes or hypertension
* Concurrent non-dietary phytoestrogens or hormone use; Vegans (vegetarians who tend to consume greater than average dose of phytoestrogens)
* Concurrent participation in other clinical trial(s)
* Unavailable for followup

Ages: 45 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30
Dates: Start 2001-02; Study Completion 2002-02

PRIMARY OUTCOMES:
safety

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Banuvar, MHSA, CCRC, Study Director — University of Illinois at Chicago

REFERENCES:
- See also: Click here for information on the UIC/NIH Center for Botanical Dietary Supplements Research — http://www.uic.edu/pharmacy/research/diet/